CLINICAL TRIAL: NCT07364604
Title: Very Early Outcomes in Endoscopic Versus Open Carpal Tunnel Release
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 64461
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Endoscopic carpal tunnel release; Open carpal tunnel release
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopic Carpal Tunnel Release: Patients who underwent endoscopic carpal tunnel release
  Interventions: Procedure: Carpal Tunnel Release
- Open Carpal Tunnel Release: Patients who underwent open carpal tunnel release
  Interventions: Procedure: Carpal Tunnel Release

INTERVENTIONS:
Procedure: Carpal Tunnel Release — Description: An open incision was made over the proximal palm to access and visualize transverse carpal tunnel, then divided it completely surgically. In the endoscopic technique, a small incision is made over the distal wrist and a camera and blade are within the wrist, then the transverse carpal ligament is divide from inside the palm

SUMMARY:
We are looking at whether there is a difference in pain and function in the very early period when comparing carpal tunnel release performed by the endoscopic technique versus the open technique.

DETAILED DESCRIPTION:
The purpose of our study is to examine the very early (<2 weeks post-op) outcomes of endoscopic versus open carpal tunnel releases (CTR). We will call patients on post-operative days 3, 7 and 14 and collect Single Assessment Numeric Evaluation (SANE), Patient Related Wrist and Hand Evaluation (PRWHE), Visual Analog Scale (VAS) pain and return to work status at each time frame to see if there is any difference between the two procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Diagnosed with carpal tunnel syndrome and indicated to undergo carpal tunnel release with one of the three participating hand surgeons were included in this study.

Exclusion Criteria:

* Patients younger than 18 years old
* Pregnant women
* Revision carpal tunnel surgery, or patients who underwent any other type of surgery concomitantly with the carpal tunnel release.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older, diagnosed with carpal tunnel syndrome and indicated to undergo carpal tunnel release with one of the three participating hand surgeons.
  Carpal tunnel syndrome was diagnosed using the physical exam, including two-point discrimination, Phalen's test, Durkan's nerve compression test, and Tinel's sign in all study participants. All patients included in the study demonstrated a CTS-6 score over 12. An electromyography (EMG) of the median nerve was performed when determined to be necessary by either the treating surgeon or referring physician.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | This was assessed at post-operative days 3, 7, and 14
  This was evaluated by administering the Patient Related Wrist and Hand Evaluation (PRWHE) questionnaire as well as obtaining a pain score using the Visual Analog Scale (VAS).
Function | Function was assessed at post-operative days 3, 7 and 14.
  Patients were first asked to assess the function of their operative hand and wrist using the Single Assessment Numeric Evaluation (SANE) tool. Function was also assessed by administering the Patient Related Wrist and Hand Evaluation (PRWHE) questionnaire.

SECONDARY OUTCOMES:
Return to Work Status | Return to work status was assessed at post-operative days 3, 7, and 14.
  Of those study patients who were not retired, we assessed if and when patients returned to work.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Yao, MD, Principal Investigator — Stanford Department of Orthopedic Surgery; Robert J Reitz, MD, Study Director — Stanford Department of Orthopedic Surgery
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta SP, MacDermid JC, Richardson J, MacIntyre NJ, Grewal R. A systematic review of the measurement properties of the patient-rated wrist evaluation. J Orthop Sports Phys Ther. 2015 Apr;45(4):289-98. doi: 10.2519/jospt.2015.5236. PMID 25827124
- [Background] Gire JD, Koltsov JCB, Segovia NA, Kenney DE, Yao J, Ladd AL. Single Assessment Numeric Evaluation (SANE) in Hand Surgery: Does a One-Question Outcome Instrument Compare Favorably? J Hand Surg Am. 2020 Jul;45(7):589-596. doi: 10.1016/j.jhsa.2020.03.024. Epub 2020 May 29. PMID 32482496
- [Background] Kishan A, Kubsad S, Haft M, Fox HM, Tuffaha SH, LaPorte DM, Nguyen DM. Endoscopic Versus Open Treatment of Carpal Tunnel Syndrome: Postoperative Complications in Patients With Diabetes Mellitus. J Hand Surg Glob Online. 2024 Jun 12;6(4):577-582. doi: 10.1016/j.jhsg.2024.04.015. eCollection 2024 Jul. PMID 39166198
- [Background] Li Y, Luo W, Wu G, Cui S, Zhang Z, Gu X. Open versus endoscopic carpal tunnel release: a systematic review and meta-analysis of randomized controlled trials. BMC Musculoskelet Disord. 2020 Apr 27;21(1):272. doi: 10.1186/s12891-020-03306-1. PMID 32340621
- [Background] Ilyas AM, Miller AJ, Graham JG, Matzon JL. Pain Management After Carpal Tunnel Release Surgery: A Prospective Randomized Double-Blinded Trial Comparing Acetaminophen, Ibuprofen, and Oxycodone. J Hand Surg Am. 2018 Oct;43(10):913-919. doi: 10.1016/j.jhsa.2018.08.011. PMID 30286851
- [Background] Sayegh ET, Strauch RJ. Open versus endoscopic carpal tunnel release: a meta-analysis of randomized controlled trials. Clin Orthop Relat Res. 2015 Mar;473(3):1120-32. doi: 10.1007/s11999-014-3835-z. Epub 2014 Aug 19. PMID 25135849
- [Background] Atroshi I, Larsson GU, Ornstein E, Hofer M, Johnsson R, Ranstam J. Outcomes of endoscopic surgery compared with open surgery for carpal tunnel syndrome among employed patients: randomised controlled trial. BMJ. 2006 Jun 24;332(7556):1473. doi: 10.1136/bmj.38863.632789.1F. Epub 2006 Jun 15. PMID 16777857
- [Background] Saw NL, Jones S, Shepstone L, Meyer M, Chapman PG, Logan AM. Early outcome and cost-effectiveness of endoscopic versus open carpal tunnel release: a randomized prospective trial. J Hand Surg Br. 2003 Oct;28(5):444-9. doi: 10.1016/s0266-7681(03)00097-4. PMID 12954254
- [Background] Chen L, Duan X, Huang X, Lv J, Peng K, Xiang Z. Effectiveness and safety of endoscopic versus open carpal tunnel decompression. Arch Orthop Trauma Surg. 2014 Apr;134(4):585-93. doi: 10.1007/s00402-013-1898-z. Epub 2014 Jan 12. PMID 24414237
- [Background] Aslani HR, Alizadeh K, Eajazi A, Karimi A, Karimi MH, Zaferani Z, Hosseini Khameneh SM. Comparison of carpal tunnel release with three different techniques. Clin Neurol Neurosurg. 2012 Sep;114(7):965-8. doi: 10.1016/j.clineuro.2012.02.017. Epub 2012 Mar 14. PMID 22421246
- [Background] Miles MR, Shetty PN, Bhayana K, Yousaf IS, Sanghavi KK, Giladi AM. Early Outcomes of Endoscopic Versus Open Carpal Tunnel Release. J Hand Surg Am. 2021 Oct;46(10):868-876. doi: 10.1016/j.jhsa.2021.04.030. Epub 2021 May 25. PMID 34049728
- [Background] Macdermid JC, Richards RS, Roth JH, Ross DC, King GJ. Endoscopic versus open carpal tunnel release: a randomized trial. J Hand Surg Am. 2003 May;28(3):475-80. doi: 10.1053/jhsu.2003.50080. PMID 12772108
- [Background] Agee JM, McCarroll HR Jr, Tortosa RD, Berry DA, Szabo RM, Peimer CA. Endoscopic release of the carpal tunnel: a randomized prospective multicenter study. J Hand Surg Am. 1992 Nov;17(6):987-95. doi: 10.1016/s0363-5023(09)91044-9. PMID 1430964
- [Background] Graham B. The value added by electrodiagnostic testing in the diagnosis of carpal tunnel syndrome. J Bone Joint Surg Am. 2008 Dec;90(12):2587-93. doi: 10.2106/JBJS.G.01362. PMID 19047703
- [Background] Williamson ERC, Vasquez Montes D, Melamed E. Multistate Comparison of Cost, Trends, and Complications in Open Versus Endoscopic Carpal Tunnel Release. Hand (N Y). 2021 Jan;16(1):25-31. doi: 10.1177/1558944719837020. Epub 2019 Mar 29. PMID 30924367
- [Background] Barnes JI, Paci G, Zhuang T, Baker LC, Asch SM, Kamal RN. Cost-Effectiveness of Open Versus Endoscopic Carpal Tunnel Release. J Bone Joint Surg Am. 2021 Feb 17;103(4):343-355. doi: 10.2106/JBJS.19.01354. PMID 33591684
- [Background] Vasiliadis HS, Georgoulas P, Shrier I, Salanti G, Scholten RJ. Endoscopic release for carpal tunnel syndrome. Cochrane Database Syst Rev. 2014 Jan 31;2014(1):CD008265. doi: 10.1002/14651858.CD008265.pub2. PMID 24482073
- [Background] Trumble TE, Diao E, Abrams RA, Gilbert-Anderson MM. Single-portal endoscopic carpal tunnel release compared with open release : a prospective, randomized trial. J Bone Joint Surg Am. 2002 Jul;84(7):1107-15. doi: 10.2106/00004623-200207000-00003. PMID 12107308
- [Background] Okutsu I, Ninomiya S, Takatori Y, Ugawa Y. Endoscopic management of carpal tunnel syndrome. Arthroscopy. 1989;5(1):11-8. doi: 10.1016/0749-8063(89)90084-4. PMID 2706046
- [Background] Shin EK. Endoscopic Versus Open Carpal Tunnel Release. Curr Rev Musculoskelet Med. 2019 Dec;12(4):509-514. doi: 10.1007/s12178-019-09584-0. PMID 31773481
- [Background] Fajardo M, Kim SH, Szabo RM. Incidence of carpal tunnel release: trends and implications within the United States ambulatory care setting. J Hand Surg Am. 2012 Aug;37(8):1599-605. doi: 10.1016/j.jhsa.2012.04.035. Epub 2012 Jun 23. PMID 22727925